CLINICAL TRIAL: NCT00793715
Title: Decompressive Laparotomy With Temporary Abdominal Closure Versus Percutaneous Puncture With Placement of Abdominal Catheter in Patients With Abdominal Compartment Syndrome During Acute Pancreatitis:Multicenter, Randomised, Controlled Study
Brief Title: Laparotomy Versus Percutaneous Puncture in Patients With Abdominal Compartment Syndrome During Acute Pancreatitis
Acronym: DECOMPRESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Belgrade (Other)
Responsible Party: Dr Dejan Radenkovic, Clinical Center of Serbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H231
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-06

CONDITIONS: Mortality; Acute Pancreatitis
Keywords: acute pancreatitis; abdominal compartment syndrome; decompressive laparotomy; percutaneous abdominal puncture; Mortality of patients treated in both arms
MeSH Terms: conditions — Pancreatitis; Intra-Abdominal Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Decompressive laparotomy with temporary abdominal closure
  Interventions: Procedure: Decompressive laparotomy with temporary abdominal closure
- 2 (Active Comparator): Patients who will receive percutaneous puncture with placement of abdominal catheter
  Interventions: Procedure: Percutaneous puncture with placement of abdominal catheter

INTERVENTIONS:
Procedure: Decompressive laparotomy with temporary abdominal closure — Surgical intervention including midline incision with temporary abdominal closure and several planed staged relaparotomies
  Arms: 1
Procedure: Percutaneous puncture with placement of abdominal catheter — Installation of abdominal catheter percutaneously via abdominal centesis 2cm bellow the umbilicus
  Arms: 2

SUMMARY:
Decompressive laparotomy with temporary abdominal closure, will decrease of overall mortality and major morbidity in patients with abdominal compartment syndrome during acute pancreatitis in comparison with percutaneous puncture with placement of abdominal catheter.

DETAILED DESCRIPTION:
We anticipated that decompressive laparotomy with temporary abdominal closure, beside all potentially negative side effects that early open surgery carries in patients with acute pancreatitis, results in decrease of overall mortality and major morbidity. The DECOMPRESS study is designed to compare effects of decompressive laparotomy with temporary abdominal closure and percutaneous puncture with placement of abdominal catheter in patients with abdominal compartment syndrome during acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* The study population consists of patients with acute pancreatitis complicated with development of abdominal compartment syndrome.

Exclusion Criteria:

* Patients will not be enrolled to the study if any of the following criteria will be present:

  * age < 18 and > 80 years
  * recent surgical interventions
  * psychoses
  * pregnancy
  * previously history of chronic pancreatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Mortality rate during the hospital stay for patients with abdominal compartment syndrome during acute pancreatitis. | 2 years

SECONDARY OUTCOMES:
duration time of organ failure | 2 years
development of a new organ failure | 2 years
number of infectious complications, | 2 years
needs for necrosectomy, | 2 years
intensive care stay | 2 years
total hospital stay | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dejan V Radenkovic, MD, PhD, Principal Investigator — Clinic for Emergency Surgery, Clinical Center of Serbia and School of Medicine, and University of Belgrade
Locations (5):
- Serbia (5):
  - Clinic for Emergency Surgery, Clinical Center of Serbia and School of Medicine, University of Belgrade, Belgrade
  - Surgical Department, Clinical Center "Bezanijska Kosa" and School of Medicine, University of Belgrade, Belgrade
  - Surgical Department, Clinical Center "Zvezdara" and School of Medicine, University of Belgrade, Belgrade
  - Surgical Department, Military-Medical Academy, Belgrade
  - Surgical Department, Clinical Center "Dr Dragisa Misovic," and School of Medicine, University of Belgrade,, Belgrade

REFERENCES:
- [Derived] Radenkovic DV, Bajec D, Ivancevic N, Bumbasirevic V, Milic N, Jeremic V, Gregoric P, Karamarkovic A, Karadzic B, Mirkovic D, Bilanovic D, Scepanovic R, Cijan V. Decompressive laparotomy with temporary abdominal closure versus percutaneous puncture with placement of abdominal catheter in patients with abdominal compartment syndrome during acute pancreatitis: background and design of multicenter, randomised, controlled study. BMC Surg. 2010 Jul 12;10:22. doi: 10.1186/1471-2482-10-22. PMID 20624281